CLINICAL TRIAL: NCT02231398
Title: Pregnancy as a Window to Future Cardiovascular Health: Adverse Pregnancy Outcomes as Predictors of Increased Risk Factors for Cardiovascular Disease
Brief Title: nuMoM2b Heart Health Study
Acronym: nuMoM2b-HHS
Status: Completed | Type: Observational
Sponsor: RTI International (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Becky McNeil, Senior Research Statistician, RTI International
Other Study IDs: NHLBI-nuMoM2b-HHS-001; 1U10HL119991 (NIH)
Record Dates: First submitted 2014-08-28; First posted 2014-09-04 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Pregnancy Complicated by Cardiovascular Disorders as Postpartum Condition, Delivered During Previous Episode; Breathing-Related Sleep Disorder
Keywords: Cardiovascular disease; Pregnant women; Nulliparity; Pregnancy outcomes; Pregnancy complications; Sleep disordered breathing
MeSH Terms: conditions — Cardiovascular Diseases; Pregnancy Complications; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples: A research or clinical staff member collects a fasting blood draw from the participant: 2 SST (tiger top) 10 mL tubes for serum; 2 EDTA (purple top) 10 mL tubes for plasma, and 1 (light blue top) 2.7 mL tube for citrated plasma. Less than 3 tablespoons of blood are collected. A 0.5 mL aliquot of whole blood from the EDTA tube is reserved. The rest of the blood is processed and as many 0.5 mL aliquots of serum, EDTA plasma, and citrated plasma as possible are collected. In addition, a 1.5 mL aliquot of buffy coat is collected from one of the EDTA tubes.
  Urine Sample: A research or clinical staff member collects about 20 mL of clean catch urine from the participant and 2 urine aliquots (1.8 mL each).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women who participated in nuMoM2b

SUMMARY:
This study is looking at the relationship between experiences during pregnancy and cardiovascular health 2 to 3½ years later. The investigators are recruiting women from the approximately 10,000 women who were enrolled and followed over the course of their first pregnancy in another study.

DETAILED DESCRIPTION:
The National Heart, Lung, and Blood Institute (NHLBI), in collaboration with the Eunice Kennedy Shriver National Institute of Child Health and Human Development, is funding this follow-up study of the nuMoM2b cohort to evaluate the association between adverse pregnancy outcomes (APOs) and cardiovascular health approximately 2 to 3½ years postpartum. The study, called the nuMoM2b Heart Health Study or nuMoM2b HHS, utilizes the extensive database and tissue bank developed for nuMoM2b in which nulliparous women are evaluated over the course of pregnancy to study the mechanisms for and prediction of APOs. Women enrolled in the nuMoM2b cohort are extremely well phenotyped through prospective data collection, clinical evaluations, and ultrasound assessments, as well as through the use of standardized definitions. Demographic, psychosocial, dietary, physiologic, and outcome information were collected through maternal interviews, self-administered questionnaires, clinical measurements, ultrasounds, and medical record abstraction. Samples of maternal blood, urine, and cervico-vaginal fluid over pregnancy and cord blood and placenta at delivery were collected and banked. All women completed two sleep questionnaires and over 3,600 had objective overnight sleep studies at two times during pregnancy.

Women participating in the nuMoM2b are assessed in nuMoM2b HHS for evidence of cardiovascular disease risk (CVDR), including sleep disordered breathing (SDB), at 2 to 3½ years postpartum. APOs in subsequent pregnancies also are assessed. This study characterizes the relationship between APOs and CVDR, identify first pregnancy profiles that portend subsequent CVDR, determine associations between SDB during the first pregnancy and subsequent CVDR, and identify modifiable factors that mediate the associations between CVDR and APOs in the first and subsequent pregnancy. This follow-up study will allow for the development of strategies to modify these CVDR factors and to improve the health of women suffering APOs.

The nuMoM2b Heart Health Study is a prospective observational study that includes interval contacts and a detailed cardiovascular assessment 2 to 3½ years after delivery of the index pregnancy. At the cardiovascular assessment, potentially eligible women are invited to attend a cardiovascular screening visit. After informed consent, a urine pregnancy test is performed to confirm eligibility. The visit includes clinical and laboratory measurements as well as a structured interview to assess domains that were measured in the nuMoM2b pregnancy: physical activity, depression, social support, psychological stress, and nutritional status. Women with sleep breathing assessments during their nuMoM2b pregnancy are offered another overnight sleep study.

The overarching goal is to better define the relation between outcomes of pregnancy and long term health of the mother. The specific aims are as follows:

Aim 1: Define the incidence of hypertension and the cardiovascular disease risk (CVDR) profile of women approximately 2 to 3½ years after a first pregnancy complicated by preeclampsia or other adverse pregnancy outcomes (APOs: stillbirth, small for gestational age at birth [SGA], preterm birth, preeclampsia, pregnancy-associated hypertension, gestational diabetes [GDM]) compared to women having no APOs in the first pregnancy.

Aim 2: Identify a profile in early pregnancy that portends subsequent CVDR approximately 2 to 3½ years postpartum.

Aim 3: Determine whether pregnancy and postpartum sleep disordered breathing (SDB) is associated with increased CVDR and identify specific patterns of pregnancy and postpartum SDB that increase CVDR.

Aim 4: Identify modifiable factors during and after pregnancy that mediate the associations between APOs and the CVDR during pregnancy and approximately 2 to 3½ years postpartum.

ELIGIBILITY:
Inclusion Criteria:

Interval Contact:

* Agreed to contact for future studies during nuMoM2b and not subsequently withdrawn from the cohort.
* Have pregnancy outcome data from the nuMoM2b study.
* At least 18 years of age (to begin interval contact attempts once nuMoM2b participant reaches age 18).
* Provision of verbal consent for telephone interview or acknowledgement of consent with completion of the web-based self-administered questionnaire.

In-clinic Visit:

* Consented for participation in interval contacts and not subsequently withdrawn
* Between 2 and 3.5 years after the nuMoM2b pregnancy ended
* Self-report at least 6 months postpartum from any subsequent pregnancy
* Self-report not currently pregnant
* Able to provide informed consent
* Provision of written, signed, informed consent for the 2 to 3.5 year in-clinic assessment
* Not currently pregnant by urine pregnancy test administered in the clinic following consent

In-home Sleep Breathing Assessment after the In-Clinic Visit:

* Participation in the in-clinic visit
* Participation in the sleep breathing substudy of nuMoM2b with at least one sleep breathing assessment providing valid data
* Not currently using positive airway pressure (PAP) therapy or other approved treatments for sleep apnea such as oral appliances and nasal therapy patch (Provent)
* Not currently on continuous oral steroid therapy for 14 days or more to treat asthma
* Not currently using oxygen supplementation to treat a medical condition
* Able to provide informed consent and deemed likely to return equipment in a reasonable period
* Provision of written, signed, informed consent for the sleep breathing assessment for the nuMoM2b Heart Health Study

Exclusion Criteria:

* Inability or refusal to provide informed consent for the study component.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible women are recruited from the cohort enrolled to nuMoM2b. For nuMom2b a convenience sample was recruited through 8 primary clinical sites that NIH selected because they could each demonstrate access to more than 4,500 deliveries per year. As a group, sites were geographically dispersed and ethically diverse. All nulliparous women aged 13 years or greater with a singleton pregnancy less than 13 weeks 6 days gestation who presented at recruitment clinics or practices and planned to deliver at a study hospital were potentially eligible for participation. A clinical or research ultrasound, performed by a study certified sonographer, confirmed viability of a singleton gestation with no obvious malformations and estimated gestational age less than or equal to 13 weeks 6 days before the woman was allowed enrollment. The first visit was scheduled and completed within a window of 6 weeks 0 days and 13 weeks 6 days estimated gestational age.
Sampling Method: Non-Probability Sample
Enrollment: 4509 (Actual)
Dates: Start 2014-09; Primary Completion 2017-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Hypertension, defined as systolic blood pressure above 140 mm Hg or diastolic blood pressure above 90 mm Hg | Blood pressures taken at study clinic visit between 2 and 3.5 years postpartum
  Will exclude participants with chronic hypertension or pregestational diabetes during or just prior to the index pregnancy.

SECONDARY OUTCOMES:
Systolic blood pressure in mm Hg | Blood pressures taken at study clinic visit between 2 and 3.5 years postpartum
  Will exclude participants with chronic hypertension or pregestational diabetes during or just prior to the index pregnancy.
Diastolic blood pressures in mm Hg | Blood pressures taken at study clinic visit between 2 and 3.5 years postpartum
  Will exclude participants with chronic hypertension or pregestational diabetes during or just prior to the index pregnancy.
HDL cholesterol in mg/dL from blood sample following overnight fast of at least 8 hours | Blood sample taken at study clinic visit between 2 and 3.5 years postpartum
  Will exclude participants with chronic hypertension or pregestational diabetes during or just prior to the index pregnancy.
LDL cholesterol in mg/dL from blood sample following overnight fast of at least 8 hours | Blood sample taken at study clinic visit between 2 and 3.5 years postpartum
  Will exclude participants with chronic hypertension or pregestational diabetes during or just prior to the index pregnancy.
Triglycerides in mg/dL from blood sample following overnight fast of at least 8 hours | Blood sample taken at study clinic visit between 2 and 3.5 years postpartum
  Will exclude participants with chronic hypertension or pregestational diabetes during or just prior to the index pregnancy.
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) from glucose and insulin measured from blood sample following overnight fast of at least 8 hours | Blood sample taken at study clinic visit between 2 and 3.5 years postpartum
  Will exclude participants with chronic hypertension or pregestational diabetes during or just prior to the index pregnancy.
High sensitivity C-reactive protein (hs-CRP) in mg/L measured from blood sample following overnight fast of at least 8 hours | Taken at study clinic visit between 2 and 3.5 years postpartum
  Will exclude participants with chronic hypertension or pregestational diabetes during or just prior to the index pregnancy.
Hemoglobin A1c (%) measured from blood sample following overnight fast of at least 8 hours | Taken at study clinic visit between 2 and 3.5 years postpartum
  Will exclude participants with chronic hypertension or pregestational diabetes during or just prior to the index pregnancy.
Sleep disordered breathing, defined as apnea-hypopnea index (AHI) of 3 or more | Taken at study clinic visit between 2 and 3.5 years postpartum
  AHI calculated for apnea-hypopnea events with 3% desaturation.

OTHER OUTCOMES:
N-terminal of the Prohormone Brain Natriuretic peptide (NT-proBNP) in pg/mL from blood sample following overnight fast of at least 8 hours | Blood sample taken at study clinic visit between 2 and 3.5 years postpartum
  project funds permitting

CONTACTS AND LOCATIONS:
Overall Officials: George Saade, M.D., Study Chair — The University of Texas Medical Branch, Galveston; Brian M. Mercer, MD, Principal Investigator — Case Western Reserve University; Ronald Wapner, MD, Principal Investigator — Columbia University; David M. Haas, M.D., M.S.,, Principal Investigator — Indiana University; Hyagriv N. Simhan, MD, MSCR, Principal Investigator — Magee Womens Hospital - University of Pittsburgh; William Grobman, M.D., M.B.A., Principal Investigator — Northwestern University; Judith Chung, M.D., Principal Investigator — University CA Irvine; Samuel Parry, M.D., Principal Investigator — University of Pennsylvania; Robert M. Silver, M.D., Principal Investigator — University of Utah
Locations (15):
- United States (15):
  - Fountain Valley Regional Hospital and Medical Center- UCI MFM private practice, Fountain Valley, California
  - Long Beach Memorial Medical Center, Women's and Children's Hospital - Women's Perinatal Group, OB Clinic, Long Beach, California
  - University of California, Irvine, Medical Center - Prenatal care clinics and private practice, Orange, California
  - Christiana Care Health Systems, Newark, Delaware
  - Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine OB/GYN, Indianapolis, Indiana
  - Columbia University Medical Center- Department of OB/GYN Division of Maternal Fetal Medicine, New York, New York
  - Case Western Reserve University, MetroHealth Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - McKay Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - University of Utah, Salt Lake City, Utah
  - Intermountain Medical Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available through an NIH data repository.

REFERENCES:
- [Background] Haas DM, Ehrenthal DB, Koch MA, Catov JM, Barnes SE, Facco F, Parker CB, Mercer BM, Bairey-Merz CN, Silver RM, Wapner RJ, Simhan HN, Hoffman MK, Grobman WA, Greenland P, Wing DA, Saade GR, Parry S, Zee PC, Reddy UM, Pemberton VL, Burwen DR; National Heart, Lung, and Blood Institute nuMoM2b Heart Health Study Network. Pregnancy as a Window to Future Cardiovascular Health: Design and Implementation of the nuMoM2b Heart Health Study. Am J Epidemiol. 2016 Mar 15;183(6):519-30. doi: 10.1093/aje/kwv309. Epub 2016 Jan 28. PMID 26825925
- [Background] Catov JM, Parker CB, Gibbs BB, Bann CM, Carper B, Silver RM, Simhan HN, Parry S, Chung JH, Haas DM, Wapner RJ, Saade GR, Mercer BM, Bairey-Merz CN, Greenland P, Ehrenthal DB, Barnes SE, Shanks AL, Reddy UM, Grobman WA; NICHD NuMoM2b and NHLBI NuMoM2b Heart Health Study Network. Patterns of leisure-time physical activity across pregnancy and adverse pregnancy outcomes. Int J Behav Nutr Phys Act. 2018 Jul 11;15(1):68. doi: 10.1186/s12966-018-0701-5. PMID 29996930
- [Background] Facco FL, Parker CB, Hunter S, Reid KJ, Zee PC, Silver RM, Haas DM, Chung JH, Pien GW, Nhan-Chang CL, Simhan HN, Parry S, Wapner RJ, Saade GR, Mercer BM, Torres C, Knight J, Reddy UM, Grobman WA; NICHD NuMoM2b and NHLBI NuMoM2b Heart Health Study Networks. Association of Adverse Pregnancy Outcomes With Self-Reported Measures of Sleep Duration and Timing in Women Who Are Nulliparous. J Clin Sleep Med. 2018 Dec 15;14(12):2047-2056. doi: 10.5664/jcsm.7534. PMID 30518449
- [Derived] Haas DM, Yang Z, Parker CB, Chung J, Parry S, Grobman WA, Mercer BM, Simhan HN, Silver RM, Wapner RJ, Saade GR, Greenland P, Merz NB, Reddy UM, Pemberton VL; nuMoM2b study and the nuMoM2b Heart Health Study. Factors associated with duration of breastfeeding in women giving birth for the first time. BMC Pregnancy Childbirth. 2022 Sep 22;22(1):722. doi: 10.1186/s12884-022-05038-7. PMID 36138368
- [Derived] Facco FL, Redline S, Hunter SM, Zee PC, Grobman WA, Silver RM, Louis JM, Pien GW, Mercer B, Chung JH, Bairey Merz CN, Haas DM, Nhan-Chang CL, Simhan HN, Schubert FP, Parry S, Reddy U, Saade GR, Hoffman MK, Levine LD, Wapner RJ, Catov JM, Parker CB. Sleep-disordered Breathing in Pregnancy and after Delivery: Associations with Cardiometabolic Health. Am J Respir Crit Care Med. 2022 May 15;205(10):1202-1213. doi: 10.1164/rccm.202104-0971OC. PMID 35144521
- [Derived] Hawkins M, Parker CB, Redline S, Larkin JC, Zee PP, Grobman WA, Silver RM, Louis JM, Pien GW, Basner RC, Chung JH, Haas DM, Nhan-Chang CL, Simhan HN, Blue NR, Parry S, Reddy U, Facco F; NICHD NuMoM2b and NHLBI NuMoM2b Heart Health Study Networks. Objectively assessed sleep-disordered breathing during pregnancy and infant birthweight. Sleep Med. 2021 May;81:312-318. doi: 10.1016/j.sleep.2021.02.043. Epub 2021 Feb 27. PMID 33756281
- [Derived] Catov JM, McNeil RB, Marsh DJ, Mercer BM, Bairey Merz CN, Parker CB, Pemberton VL, Saade GR, Chen YI, Chung JH, Ehrenthal DB, Grobman WA, Haas DM, Parry S, Polito L, Reddy UM, Silver RM, Simhan HN, Wapner RJ, Kominiarek M, Kreutz R, Levine LD, Greenland P; NHLBI nuMoM2b Heart Health Study. Early Pregnancy Atherogenic Profile in a First Pregnancy and Hypertension Risk 2 to 7 Years After Delivery. J Am Heart Assoc. 2021 Feb;10(5):e017216. doi: 10.1161/JAHA.120.017216. Epub 2021 Feb 23. PMID 33619977
- [Derived] Haas DM, Parker CB, Marsh DJ, Grobman WA, Ehrenthal DB, Greenland P, Bairey Merz CN, Pemberton VL, Silver RM, Barnes S, McNeil RB, Cleary K, Reddy UM, Chung JH, Parry S, Theilen LH, Blumenthal EA, Levine LD, Mercer BM, Simhan H, Polito L, Wapner RJ, Catov J, Chen I, Saade GR; NHLBI nuMoM2b Heart Health Study. Association of Adverse Pregnancy Outcomes With Hypertension 2 to 7 Years Postpartum. J Am Heart Assoc. 2019 Oct;8(19):e013092. doi: 10.1161/JAHA.119.013092. Epub 2019 Sep 30. PMID 31564189
- [Derived] Monk C, Webster RS, McNeil RB, Parker CB, Catov JM, Greenland P, Bairey Merz CN, Silver RM, Simhan HN, Ehrenthal DB, Chung JH, Haas DM, Mercer BM, Parry S, Polito L, Reddy UM, Saade GR, Grobman WA; NICHD nuMoM2b and NHLBI nuMoM2b Heart Health Study Networks. Associations of perceived prenatal stress and adverse pregnancy outcomes with perceived stress years after delivery. Arch Womens Ment Health. 2020 Jun;23(3):361-369. doi: 10.1007/s00737-019-00970-8. Epub 2019 Jun 29. PMID 31256258